CLINICAL TRIAL: NCT01695252
Title: Measuring and Monitoring Patient Informed Clinical Outcomes In Psychological Therapy Supervision - A Stepped Wedge Cluster Randomised Controlled Trial
Brief Title: Measuring and Monitoring Patient Informed Clinical Outcomes In Psychological Therapy Supervision
Acronym: MEMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Professor Kate Davidson, Director of Glasgow Institute of Psychological Interventions, NHS Greater Glasgow and Clyde
Allocation: Randomized | Purpose: Treatment
Other Study IDs: GN12CP071; CZH/4/708 (Other Grant/Funding Number: Chief Scientist Office)
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Patients Referred for Routine Psychological Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-Sup (No Intervention): Standard supervision
- MEMOS (Experimental): Patient informed clinical outcomes supervision
  Interventions: Other: MEMOS

INTERVENTIONS:
Other: MEMOS — Patient informed clinical outcomes supervision
  Arms: MEMOS

SUMMARY:
Providing feedback on patient progress to therapists improves clinical outcomes for patients, particularly those who are failing to improve with therapy. The encouraging research has been carried out by a small group of researchers, largely working in the United States health care context. The samples studied have been young people attending university counselling services, suffering from mild mental health disorders. The group studies are therefore not similar to patients seen for psychological therapy in the NHS. Also given that therapists are not necessarily alert to treatment failure, have an overly optimistic view of their patients progress even when provided with evidence to the contrary, clinical supervision may be a more effective method through which to provide patient informed clinical outcomes than directly to therapists themselves.

We will assess if providing feedback through the supervision process is more effective than providing this information to therapists themselves in terms of improving clinical outcomes, particularly for patients who are failing to improve with routine NHS Psychological therapy.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

Patients

Able to give informed consent Male or female (>18 years of age) Requiring psychological treatment or therapy in routine Mental Health Services Able and competent to understand and complete CORE questionnaires

Supervisors and their therapists

Able to give written informed consent Any NHS Greater Glasgow and Clyde applied psychologist who is supervising therapists offering routine psychological therapy to patients in NHS Greater Glasgow and Clyde and whose therapists agree to take part in the study.

Exclusion Criteria:

Patients

Below the age of 18 years Inability to give written informed consent Inability to understand and complete CORE questionnaires

Supervisors and their therapists

Those supervisors and therapists who are unlikely to be able to stay in the study for its duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Overall CORE-OM score
  Change from baseline at discharge and 6 months follow-up in the primary outcome will be compared between the supervision groups using a repeated measure analysis with appropriate correlation structure, including a random effect for therapist and fixed effects for baseline overall CORE-OM score and any other appropriate demographics.

SECONDARY OUTCOMES:
CORE 10

CONTACTS AND LOCATIONS:
Overall Officials: Kate M Davidson, MA MPhil PhD, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

REFERENCES:
- [Background] Davidson KM, Rankin ML, Begley A, Lloyd S, Barry SJ, McSkimming P, Bell L, Allan C, Osborne M, Ralston G, Bienkowski G, Mellor-Clark J, Walker A. Assessing Patient Progress in Psychological Therapy Through Feedback in Supervision: the MeMOS* Randomized Controlled Trial (*Measuring and Monitoring clinical Outcomes in Supervision: MeMOS). Behav Cogn Psychother. 2017 May;45(3):209-224. doi: 10.1017/S1352465817000029. Epub 2017 Feb 7. PMID 28166849